CLINICAL TRIAL: NCT02508714
Title: Bioresorbable Polymer ORSIRO Versus Durable Polymer RESOLUTE ONYX Stents (BIONYX): A Randomized Trial With Stent Evaluation in All-comers IV (TWENTE IV)
Brief Title: Bioresorbable Polymer ORSIRO Versus Durable Polymer RESOLUTE ONYX Stents
Acronym: BIONYX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Thorax Centrum Twente (Other)
Responsible Party: Principal Investigator, Clemens von Birgelen, MD, PhD, Thorax Centrum Twente
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P15-19
Record Dates: First submitted 2015-07-23; First posted 2015-07-27 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: Coronary Artery Disease; Angina Pectoris; Unstable Angina Pectoris; Acute Coronary Syndrome; Coronary Stenosis; Coronary Restenosis
MeSH Terms: conditions — Coronary Artery Disease; Angina Pectoris; Angina, Unstable; Acute Coronary Syndrome; Coronary Stenosis; Coronary Restenosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Orsiro DES (Biotronik) (Active Comparator): The ORSIRO hybrid coating DES (Biotronik, Switzerland) is a device which includes a modern, highly flexible, thin-strut stent platform, eluting sirolimus from a thin biodegradable BIO-lute coating grom PLLA (poly(L-lactic acid)) which is located mainly on the abluminal side.
  Interventions: Device: Orsiro
- RESOLUTE ONYX DES (Medtronic) (Active Comparator): The RESOLUTE ONYX is a permanent polymer DES that uses a novel highly flexible metallic stent backbone with increased radiographic visibility eluting the drug zotarolimus from the BioLinx durable polymer coating. The stent platform uses corewire technology that allows the stent to have a denser core metal surrounded by outer layer of cobalt-chromium.
  Interventions: Device: Resolute Onyx

INTERVENTIONS:
Device: Orsiro — stents will be implanted in case of significant coronary artery disease
  Other Names: Orsiro drug eluting stent
  Arms: Orsiro DES (Biotronik)
Device: Resolute Onyx — stents will be implanted in case of significant coronary artery disease based on coronary angiography
  Other Names: Resolute Onyx drug eluting stent
  Arms: RESOLUTE ONYX DES (Medtronic)

SUMMARY:
The introduction of drug-eluting stents (DES) in the treatment of coronary artery disease has led to a significant reduction in morbidity. However, the first generation of these devices had no positive impact on the mortality after PCI (compared to bare metal stents), which was greatly attributed to a somewhat increased incidence of late and very late stent thrombosis. Concerns about the role of durable polymers as a potential trigger of inflammation and finally adverse events also led to the development of DES with bioresorbable coatings, which leave after degradation of the coating only a bare metal stent in the vessel wall that does not induce an inflammatory response. While such bioresorbable polymer DES are increasingly used in clinical practice, data from head-to-head comparisons between bioresorbable polymer DES with a contemporary highly flexible new generation permanent polymer coated DES.

DETAILED DESCRIPTION:
rationale: The introduction of drug-eluting stents (DES) in the treatment of coronary artery disease has led to a significant reduction in morbidity. However, the first generation of these devices had no positive impact on the mortality after PCI (compared to bare metal stents), which was greatly attributed to a somewhat increased incidence of late and very late stent thrombosis. Concerns about the role of durable polymers as a potential trigger of inflammation and finally adverse events also led to the development of DES with bioresorbable coatings, which leave after degradation of the coating only a bare metal stent in the vessel wall that does not induce an inflammatory response. While such bioresorbable polymer DES are increasingly used in clinical practice, data from head-to-head comparisons between bioresorbable polymer DES with a contemporary highly flexible new generation permanent polymer coated DES.

Aim:

The aim of the study is to compare the outcome of the bioresorbable polymer coated stent (ORSIRO) and a new generation permanent polymer coated stent (RESOLUTE ONYX) in an all-comers patient population and non-inferiority setting.

Study design:

The study is a prospective, randomized, single-blinded, multicentre trial with 1:1 randomization for drug-eluting stent type, stratified for gender and the presence of diabetes mellitus.

Study population:

Patients who require percutaneous coronary intervention (PCI) for the treatment of coronary stenoses with an indication for DES use, according to current guidelines and/or the operators clinical judgement. All clinical syndromes will be included. A total of 2,470 patients will be included.

Intervention:

One group will receive the ORSIRO stent, the other group will receive the RESOLUTE ONYX stent. All other intervention and procedural characteristics are similar.

Primary study outcome:

Incidence of target vessel failure (TVF) at 1 year follow-up (according to ARC definitions). Components of the primary endpoint in hierarchical order: - Cardiac death: all deaths are considered cardiac, unless an unequivocal non-cardiac cause can be established. - Target vessel related myocardial infarction (MI) that is Q-wave or non-Q-wave, that can be related to the target vessel or cannot be related to another vessel. - Clinically driven repeated target vessel revascularization by means of PCI or coronary artery bypass grafting (CABG).

ELIGIBILITY:
Inclusion Criteria:

* Patients of 18 years and older, requiring PCI for the treatment of significant coronary artery or bypass graft lesions, being eligible for treatment with drug eluting stents according to clinical guidelines and/or the operators' judgement, and capable of providing informed consent.
* Patients with all clinical syndromes will be enrolled without any exclusion based on number, type, location or length of lesions to be treated.

Exclusion Criteria:

* Known intolerance to components of one of the study DES, or known intolerance to antithrombotic and/or anticoagulant therapy that prevents adherence to any dual anti-platelet therapy (DAPT).
* Planned elective surgical procedure necessitating interruption of DAPT during the first 3 months after randomization.
* Participation in another randomized cardiovascular device trial or randomized pharmacological study related to antithrombotic and/or anticoagulant therapy before reaching the primary endpoint.
* Known pregnancy, adherence to scheduled follow-up is unlikely, or life expectancy is assumed to be less than 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2470 (Actual)
Dates: Start 2016-10-07 (Actual); Primary Completion 2018-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Target vessel failure (TVF) | 1 year
  Composite endpoint consisting of: Cardiac death (All deaths are considered cardiac, unless an unequivocal non-cardiac cause can be established); Target vessel related MI (Q-wave or non-Q-wave myocardial infarction that can be related to the target vessel or cannot be related to another vessel); Clinically driven repeated target vessel revascularization by means of CABG or PCI.

SECONDARY OUTCOMES:
Death at 1 and 2 year follow-up | 1 and 2 year
  Death distinguished into: cardiac, vascular, other causes, all-cause mortality
Myocardial infarction at 1 and 2 year follow-up | 1 and 2 year
  Myocardial infarction distinguished into Q-wave and non-Q-wave myocardial infarction
Revascularization at 1 and 2 year follow-up | 1 and 2 year
  Target-vessel revascularization distinguished into PCI or CABG
Stent thrombosis at 1 and 2 year follow-up | 1 and 2 year
  Stent thrombosis was distinguished into definite, probable and possible according to the Academic Research Consortium (ARC) definition.
Target lesion failure (TLF) at 1 and 2 year follow-up | 1 and 2 year
  Composite endpoint consisting of : cardiac death; target vessel-related MI; clinically driven target lesion revascularization (TLR)
Major adverse cardiac events (MACE) at 1 and 2 year follow-up | 1 and 2 year follow-up
  Composite endpoint consisting of:
  1. any death;
  2. any myocardial infarction
  3. emergent CABG;
  4. clinically indicated TLR
Patient oriented composite endpoint (POCE) at 1 and 2 year follow-up | 1 and 2 year follow-up
  Composite endpoint consisting of: any death; any myocardial infarction; any revascularization.
Major Bleeding at 1 and 2 year follow-up | 1 and 2 year follow-up
  Major bleeding that require surgery or blood transfusions or cerebral hemorrhages

OTHER OUTCOMES:
Longitudinal stent deformation (LSD) and deliverability | 1 year
  Identification of deformation of a stent in the longitudinal axis during coronary angiographic assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Clemens von Birgelen, MD, PhD, Principal Investigator — Thorax Centrum Twente
Locations (7):
- Belgium (2):
  - CHU Charleroi, Charleroi
  - Jessa Ziekenhuis, Hasselt
- Rambam, Haifa, Israel
- Netherlands (4):
  - Haga Ziekenhuis, The Hague, South Holland
  - Rijnstate Hospital, Arnhem
  - Treant Zorggroep, Emmen
  - Medisch Spectrum Twente, Enschede

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] von Birgelen C, Sen H, Lam MK, Danse PW, Jessurun GA, Hautvast RW, van Houwelingen GK, Schramm AR, Gin RM, Louwerenburg JW, de Man FH, Stoel MG, Lowik MM, Linssen GC, Said SA, Nienhuis MB, Verhorst PM, Basalus MW, Doggen CJ, Tandjung K. Third-generation zotarolimus-eluting and everolimus-eluting stents in all-comer patients requiring a percutaneous coronary intervention (DUTCH PEERS): a randomised, single-blind, multicentre, non-inferiority trial. Lancet. 2014 Feb 1;383(9915):413-23. doi: 10.1016/S0140-6736(13)62037-1. Epub 2013 Oct 31. PMID 24183564
- [Background] Sen H, Lam MK, Lowik MM, Danse PW, Jessurun GA, van Houwelingen KG, Anthonio RL, Tjon Joe Gin RM, Hautvast RW, Louwerenburg JH, de Man FH, Stoel MG, van der Heijden LC, Linssen GC, IJzerman MJ, Tandjung K, Doggen CJ, von Birgelen C. Clinical Events and Patient-Reported Chest Pain in All-Comers Treated With Resolute Integrity and Promus Element Stents: 2-Year Follow-Up of the DUTCH PEERS (DUrable Polymer-Based STent CHallenge of Promus ElemEnt Versus ReSolute Integrity) Randomized Trial (TWENTE II). JACC Cardiovasc Interv. 2015 Jun;8(7):889-99. doi: 10.1016/j.jcin.2015.01.033. Epub 2015 May 20. PMID 26003019
- [Derived] van Vliet D, Pinxterhuis TH, Ploumen EH, Kok MM, Buiten RA, Zocca P, Roguin A, Schotborgh CE, Anthonio RL, Danse PW, Benit E, Aminian A, Doggen CJM, von Birgelen C. Impact of diabetes on three-year outcome after coronary stenting in patients with polyvascular atherosclerotic disease - a secondary analysis of the randomized TWENTE trials. Int J Cardiol Heart Vasc. 2025 Jul 6;59:101741. doi: 10.1016/j.ijcha.2025.101741. eCollection 2025 Aug. PMID 40687396
- [Derived] van Vliet D, Ploumen EH, Pinxterhuis TH, Doggen CJM, Aminian A, Schotborgh CE, Danse PW, Roguin A, Anthonio RL, Benit E, Kok MM, Linssen GCM, von Birgelen C. Elderly patients treated with Onyx versus Orsiro drug-eluting coronary stents in a randomized clinical trial with long-term follow-up. Clin Res Cardiol. 2025 Dec;114(12):1681-1691. doi: 10.1007/s00392-025-02622-7. Epub 2025 Mar 4. PMID 40035811
- [Derived] van Vliet D, Ploumen EH, Pinxterhuis TH, Buiten RA, Aminian A, Schotborgh CE, Danse PW, Roguin A, Anthonio RL, Benit E, Zocca P, Doggen CJM, von Birgelen C. Final 5-year report of BIONYX comparing the thin-composite wire-strut zotarolimus-eluting stent versus ultrathin-strut sirolimus-eluting stent. Catheter Cardiovasc Interv. 2024 Jul;104(1):1-9. doi: 10.1002/ccd.31067. Epub 2024 May 7. PMID 38713843
- [Derived] Pinxterhuis TH, Ploumen EH, Zocca P, Doggen CJM, Schotborgh CE, Anthonio RL, Roguin A, Danse PW, Benit E, Aminian A, Hartmann M, Linssen GCM, von Birgelen C. Impact of premature coronary artery disease on adverse event risk following first percutaneous coronary intervention. Front Cardiovasc Med. 2023 Sep 7;10:1160201. doi: 10.3389/fcvm.2023.1160201. eCollection 2023. PMID 37745109
- [Derived] Pinxterhuis TH, Ploumen EH, Zocca P, Doggen CJM, Schotborgh CE, Anthonio RL, Roguin A, Danse PW, Benit E, Aminian A, van Houwelingen KG, Linssen GCM, Geelkerken RH, von Birgelen C. Outcome of percutaneous coronary intervention using ultrathin-strut biodegradable polymer sirolimus-eluting versus thin-strut durable polymer zotarolimus-eluting stents in patients with comorbid peripheral arterial disease: a post-hoc analysis from two randomized trials. Cardiovasc Diagn Ther. 2023 Aug 31;13(4):673-685. doi: 10.21037/cdt-22-584. Epub 2023 Jul 24. PMID 37675090
- [Derived] Pinxterhuis TH, Ploumen EH, Doggen CJM, Hartmann M, Schotborgh CE, Anthonio RL, Roguin A, Danse PW, Benit E, Aminian A, Linssen GCM, von Birgelen C. First myocardial infarction in patients with premature coronary artery disease: insights into patient characteristics and outcome after treatment with contemporary stents. Eur Heart J Acute Cardiovasc Care. 2023 Nov 16;12(11):774-781. doi: 10.1093/ehjacc/zuad098. PMID 37619976
- [Derived] Pinxterhuis TH, Ploumen EH, Zocca P, Doggen CJM, Schotborgh CE, Anthonio RL, Roguin A, Danse PW, Benit E, Aminian A, Stoel MG, Linssen GCM, Geelkerken RH, von Birgelen C. Outcome after percutaneous coronary intervention with contemporary stents in patients with concomitant peripheral arterial disease: A patient-level pooled analysis of four randomized trials. Atherosclerosis. 2022 Aug;355:52-59. doi: 10.1016/j.atherosclerosis.2022.05.002. Epub 2022 May 20. PMID 35641327
- [Derived] Ploumen EH, Pinxterhuis TH, Zocca P, Roguin A, Anthonio RL, Schotborgh CE, Benit E, Aminian A, Danse PW, Doggen CJM, von Birgelen C, Kok MM. Impact of prediabetes and diabetes on 3-year outcome of patients treated with new-generation drug-eluting stents in two large-scale randomized clinical trials. Cardiovasc Diabetol. 2021 Oct 30;20(1):217. doi: 10.1186/s12933-021-01405-4. PMID 34717627
- [Derived] Ploumen EH, Buiten RA, Zocca P, Doggen CJ, Aminian A, Schotborgh CE, Jessurun GA, Roguin A, Danse PW, Benit E, von Birgelen C. First Report of 3-Year Clinical Outcome After Treatment With Novel Resolute Onyx Stents in the Randomized BIONYX Trial. Circ J. 2021 Oct 25;85(11):1983-1990. doi: 10.1253/circj.CJ-21-0292. Epub 2021 Jul 13. PMID 34261828
- [Derived] von Birgelen C, Zocca P, Buiten RA, Jessurun GAJ, Schotborgh CE, Roguin A, Danse PW, Benit E, Aminian A, van Houwelingen KG, Anthonio RL, Stoel MG, Somi S, Hartmann M, Linssen GCM, Doggen CJM, Kok MM. Thin composite wire strut, durable polymer-coated (Resolute Onyx) versus ultrathin cobalt-chromium strut, bioresorbable polymer-coated (Orsiro) drug-eluting stents in allcomers with coronary artery disease (BIONYX): an international, single-blind, randomised non-inferiority trial. Lancet. 2018 Oct 6;392(10154):1235-1245. doi: 10.1016/S0140-6736(18)32001-4. Epub 2018 Sep 22. PMID 30253879
- [Derived] van der Heijden LC, Kok MM, Zocca P, Jessurun GAJ, Schotborgh CE, Roguin A, Benit E, Aminian A, Danse PW, Lowik MM, Linssen GCM, van der Palen J, Doggen CJM, von Birgelen C. Bioresorbable Polymer-Coated Orsiro Versus Durable Polymer-Coated Resolute Onyx Stents (BIONYX): Rationale and design of the randomized TWENTE IV multicenter trial. Am Heart J. 2018 Apr;198:25-32. doi: 10.1016/j.ahj.2017.12.011. Epub 2017 Dec 21. PMID 29653644